CLINICAL TRIAL: NCT05587894
Title: OPtimisation of Antiviral Therapy in Immunocompromised COVID-19 Patients: a Randomized Factorial Controlled Strategy Trial: the OPTICOV Study
Brief Title: OPtimisation of Antiviral Therapy in Immunocompromised COVID-19 Patients: a Randomized Factorial Controlled Strategy Trial
Acronym: OPTICOV
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Alexandra Calmy, HIV/AIDS Unit Director, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 0176s OPTICOV; CT-2022-501408-81-01 (Registry Identifier: EMA CTIS)
Record Dates: First submitted 2022-10-17; First posted 2022-10-20 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: COVID-19; Immunodeficiency
MeSH Terms: conditions — COVID-19; Immunologic Deficiency Syndromes | interventions — nirmatrelvir and ritonavir drug combination; Ritonavir; remdesivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Nirmatrelvir/r 5 days alone (Experimental)
  Interventions: Drug: Paxlovid 5 days
- Nirmatrelvir/r 10 days alone (Experimental)
  Interventions: Drug: Paxlovid 10 days
- Nirmatrelvir/r 5 days + remdesivir s.d (Experimental)
  Interventions: Drug: Paxlovid 5 days; Drug: Veklury
- Nirmatrelvir/r 10 days + remdesivir s.d (Experimental)
  Interventions: Drug: Paxlovid 10 days; Drug: Veklury

INTERVENTIONS:
Drug: Paxlovid 5 days — Nirmatrelvir/r 300mg/100 mg bid will be given for 5 days, orally.
  Nirmatrelvir/r is a combination of two molecules: nirmatrelvir which is a protease inhibitor (against 3CL) and ritonavir which has a booster role.
  Nirmatrelvir/r (marketed by Pfizer under the brand name Paxlovid®) is indicated for the treatment of COVID-19 in adults who do not require supplemental oxygen and who are at increased risk for progressing to severe COVID-19.
  Other Names: Nirmatrevlir/ritonavir
  Arms: Nirmatrelvir/r 5 days + remdesivir s.d; Nirmatrelvir/r 5 days alone
Drug: Paxlovid 10 days — Nirmatrelvir/r 300mg/100 mg bid will be given for 10 days, orally.
  Other Names: Nirmatrevlir/ritonavir
  Arms: Nirmatrelvir/r 10 days + remdesivir s.d; Nirmatrelvir/r 10 days alone
Drug: Veklury — Remdesivir "flash", 200mg, intravenous. Remdesivir (marketed by Gilead under de brand name Veklury®) is indicated in patients with pneumonia requiring supplemental oxygen (inpatients), as well as in outpatients who are at increased risk of progressing to severe COVID-19. The mode of action characterize remdesivir as a direct-acting antiviral compound.
  Other Names: remdesivir
  Arms: Nirmatrelvir/r 10 days + remdesivir s.d; Nirmatrelvir/r 5 days + remdesivir s.d

SUMMARY:
The overall purpose of the trial is to evaluate the efficacy and safety of possible combination antiviral therapy DAA (remdesivir + nirmatrelvir/r)∞ versus the reference monotherapy (nirmatrelvir/r alone) and to assess the efficacy and safety of increasing the nirmatrelvir/r course from 5- to 10 days in immunocompromised patients diagnosed with asymptomatic or mild to moderate COVID-19.

DETAILED DESCRIPTION:
This is a randomized, controlled, factorial, superiority trial to evaluate the viral efficacy of DAA (nirmatrelvir/r) + DAA (remdesivir)∞ versus nirmatrelvir/r alone and of 5 days versus 10 days of nirmatrelvir/r in immunocompromised patients diagnosed with asymptomatic or mild to moderate COVID-19.

The primary objective is to assess whether (i) a combination antiviral therapy of two DAA (nirmatrelvir/r + remdesivir)∞ And/or (ii) an increase in nirmatrelvir/r duration from 5 to 10 days improves viral efficacy by decreasing the SARS-CoV-2 positivity rate by real time RT-PCR (CT<32) in nasopharyngeal swabs at D10.

Patients will be eligible if they are immunocompromised, have confirmed asymptomatic SARS-CoV-2 infection or mild to moderate COVID-19, regardless of symptoms onset, provided that they have no contra-indication to any of the study drugs.

A total of 256 patients will be included in France and Switzerland.

Participants not eligible for randomisation or who refuse to participate to the trial for any reason will be proposed to be included in an exploratory non comparative cohort (maximum 97 participants).

ELIGIBILITY:
Inclusion Criteria:

1. Laboratory confirmed SARS-CoV-2 infection by RT-PCR or positive antigenic test
2. Asymptomatic or mild to moderate COVID-19 (WHO progression scale <5). Patients receiving oxygen therapy for reasons other than a pulmonary COVID-19 are eligible)
3. ≥ 16 years of age;
4. Immunocompromised as defined by ≥ 1 risk factors for severe COVID-19 as assessed by the FOPH list (criteria 5: diseases/treatments leading to immune suppression)

   * Severe immunosuppression (e.g., HIV infection with CD4 + T cell count <350 / µl)
   * Neutropenia (<1000 neutrophils / µl) ≥1 week
   * Lymphocytopenia (<200 lymphocytes/µl)
   * Hereditary immunodeficiencies
   * Intake of drugs which suppress the immune system (e.g. glucocorticoids for a long time [an equivalent dose of prednisone >20 mg/day > 3 months], monoclonal antibodies, cytostatics, biological products, everolimus, mTOR inhibitors etc.) in the last 12 months
   * Active cancer under cytostatics or targeted therapy known to be immunosuppressive (e.g., platinum salts, cyclophosphamide, anthracyclines, taxanes, 5-fluorouracil, gemcitabine, purine inhibitors, proteasome inhibitors) or associated with hematologic toxicity (neutropenia, lymphopenia), for example sunitinib, imatinib, regorafenib
   * Aggressive lymphomas (all types)
   * Acute lymphatic leukemia
   * Acute myeloid leukemia
   * Acute promyelocytic leukemia
   * T prolymphocytic leukemia
   * Primary central nervous system lymphoma
   * Stem cell transplantation
   * Light chain amyloidosis
   * Chronic lymphoid leukemia
   * Multiple myeloma
   * Sickle cell disease
   * Bone marrow transplant
   * Organ transplant
   * Being on the waiting list for an organ transplant
5. Willing and able to comply with study requirements and restrictions as described in the informed consent form (ICF)
6. Enrolled in or a beneficiary of a Social Security program (State Medical Aid (AME) is not a Social Security program) or holders of health insurance
7. Participant's or its legal representative's signature of the informed consent form

Exclusion Criteria:

1. SARS-CoV-2 PCR ≥30 CT at screening
2. Hypersensitivity to study drugs (active substance(s) or excipients)
3. Body weight < 40 kg
4. AST or ALT > 5 times the upper limit
5. Cirrhosis Child-Pugh score C
6. Is taking or is anticipated to require any prohibited therapies*
7. Participation in another interventional clinical study through Day 28 with an investigational compound or device, including COVID-19 therapeutics, where the study intervention is performed in the 28 days preceding the inclusion and the 10 days after the inclusion. Investigators of the different clinical studies should agree on participant's inclusion
8. Presence of any condition for which, in the opinion of the investigator, participation would not be in participant's best interest or that could prevent, limit, or confound the protocol-specified assessments
9. Having received antiviral treatments against SARS-CoV-2 in the 14 days before the inclusion with exception of those having received one or two doses of nirmatrevir/r in the 24h preceding the inclusion in the study.
10. Pregnant or breastfeeding female

    * Study SOPs based on recommendations from the Liverpool COVID-19 interactions, French Society for Pharmacology and Therapeutics and French Speaking Transplantation society will be provided to guide investigators

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2023-04-27 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with SARS-CoV-2 viral load (threshold cicle (Ct) <32) by real-time RT-PCR in nasopharyngeal swabs at Day 10 after treatment initiation. | Day 10
  SARS-CoV-2 viral load is measured in nasopharyngeal swabs by real-time RT-PCR

SECONDARY OUTCOMES:
Percentage of patients with SARS-CoV-2 viral load (threshold cicle <32 CT) by real-time RT-PCR in nasopharyngeal swabs at Day5, Day14 and Day21 after treatment initiation | Day5, Day14 and Day21
  SARS-CoV-2 viral load is measured in nasopharyngeal swabs by real-time RT-PCR
Percentage of patients with detectable SARS-CoV-2 viremia at Day5, Day10 and Day14 | Assessed for 14 days from the date of randomisation at Day5, Day10 and Day14
  SARS-CoV-2 viremia is measured from plasma samples by real-time RT-PCR
Decrease of SARS-CoV-2 viral load measured by copies/ml by nasopharyngeal swab at Day5, Day10, Day14, Day21 and in blood samples at Day5, Day10 and Day14 comparatively to screening | Day5, Day10, Day14, Day21
  SARS-CoV-2 viral load is measured in nasopharyngeal swabs and in blood samples by real-time RT-PCR
Number of de novo emergence of mutations on nasopharyngeal RT-PCR at Day5, Day10, Day14 and Day21 comparatively to screening | Day5, Day10, Day14 and Day21
  Emergence of mutations is measured in nasopharyngeal swabs by genotyping techniques
Time to first negative SARS-CoV-2 RT-PCR (CT<32) until Day90 | Day90
  SARS-CoV-2 viral load is measured in nasopharyngeal swabs by real-time RT-PCR
Absence of ability to cultivate virus from viral cultures from nasopharyngeal swabs at Day5, Day10 and Day21 | Day5, Day10 and Day21
  Viral culture is performed from nasopharyngeal swabs samples
Percentage of patients with sustained resolution or abatement of symptoms defined as a FLU-PRO-Plus score ≤1 at Day5, Day10, Day14, Day21 and Day28 | Day5, Day10, Day14, Day21 and Day28
  FLU-PRO-Plus score is measured via an arithmetic formula
All-cause hospitalization and/or death at Day28 | Day28
  Outcome measured during patients medical follow-up
Hospitalization at Day28 | Day28
  Outcome measured during patients medical follow-up
Death at Day28 | Day28
  Outcome measured during patients medical follow-up
Rate of Post-COVID19 condition at Day90 according to the WHO October 2021 definition | Day 90
  Rate of Post-COVID19 condition at Day90 according to the WHO October 2021 definition:
  o Post COVID-19 condition occurs in individuals with a history of probable or confirmed SARS-CoV-2 infection, usually 3 months from the onset of COVID-19 with symptoms that last for at least 2 months and cannot be explained by an alternative diagnosis. Common symptoms include fatigue, shortness of breath, cognitive dysfunction but also others and generally have an impact on everyday functioning. Symptoms may be new onset following initial recovery from an acute COVID-19 episode or persist from the initial illness. Symptoms may also fluctuate or relapse over time.
Percentage of participants with an adverse event (AE) or serious adverse event (SAE) or AE leading to treatment discontinuation up to Day28 | Day 28
  Outcome measured during patients medical follow-up
Adherence to nirmatrelvir/r with patient-reported adherence and nirmatrelvir/r residual plasma dosage at Day5 and Day10 | Day5 and Day10
  Outcome measured by patient-reported adherence and drug residual dosage using dried spot (DBS)
Number of DDIs who led to dosage adjustment of other patient's drugs | Assessed up to Day 10 from randomisation
  Outcome measured during patients medical follow-up
Percentage of patients with specific retreatment patients (by antiviral antiinflammatory drugs or convalescent plasma through Day90 | Day90
  Outcome measured during patients medical follow-up
To assess the phenotypic resistance (IC50 increase) against treatment for viral strains cultured from nasopharyngeal swabs | Day5, Day10, Day14, Day21
  Outcome measured in nasopharyngeal swabs by phenotyping techniques
Immunosuppressors residual concentrations, if applicable | as needed
  Outcome measures in participants' blood samples

CONTACTS AND LOCATIONS:
Locations (18):
- France (14):
  - Saint-André Hospital, Bordeaux
  - Pellegrin Hospital, Bordeaux
  - Francois Mitterrand Hospital, Dijon
  - Croix Rousse Hospital, Lyon
  - La Colombière Hospital, Montpellier
  - Hotel Dieu Hospital, Nantes
  - Laribosière Hospital, Paris
  - Saint Antoine Hospital, Paris
  - Pitié-Salpêtrière Hospital, Paris
  - Saint Louis Hospital, Paris
  - Bichat Claude-Bernard Hospital, Paris
  - Robert Debré Hospital, Reims
  - Purpan Hospital, Toulouse
  - Tourcoing Hospital, Tourcoing
- Switzerland (4):
  - Basel University Hospital, Basel
  - University Hospitals of Geneva, Geneva
  - University Hospital CHUV, Lausanne
  - University Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: Undecided